CLINICAL TRIAL: NCT00939315
Title: Impact of Multimodal Diagnostic Assessment of Cerebral Gliomas With F-18-fluoroethyl-L-tyrosine PET/CT, F-18-fluorocholine PET/CT and Magnetic Resonance Imaging and Spectroscopy
Brief Title: Multimodal Diagnostic Assessment of Cerebral Gliomas With FET & FCH PET/CT, and Magnetic Resonance Imaging/Spectroscopy
Acronym: Gliomes-FLP
Status: Completed | Type: Observational
Sponsor: University of Lausanne Hospitals (Other)
Collaborators: Lionel Perrier Foundation (Montreux, Switzerland) (Unknown)
Responsible Party: Principal Investigator, John O. Prior, Professor and Head of Department, University of Lausanne Hospitals
Other Study IDs: 196/08; Swissmedic 2009DR3123 (Other: Swissmedic)
Record Dates: First submitted 2009-07-14; First posted 2009-07-15 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: Glioma
Keywords: Glioma, diagnosis; Imaging; Positron emission tomography; Magnetic resonance imaging; Magnetic resonance spectroscopy
MeSH Terms: conditions — Glioma; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to establish the diagnostic value of O-(2-[18F]-fluoroethyl)-L-tyrosine (FET) PET-CT, [18F]-fluorocholine (FCH) and magnetic resonance imaging (MRI) combined with magnetic resonance spectroscopy (MRS) in patients with suspected cerebral glioma using neuronavigated biopsies with histopathological analysis as reference.

DETAILED DESCRIPTION:
The objectives of the study are:

* To demonstrate if the multimodal approach, combining the morphological aspect of the MRI with the metabolic aspect of the tumor with magnetic resonance spectroscopy (MRS) and O-(2-[18F]-fluoroethyl)-L-tyrosine (FET) or 18F]-fluorocholine (FCH) PET/CTthe FCH allows to improve the location of a active metabolic tumor and its impact on the ideal choice of sampling biopsy.
* To underline the differences and similarities between MRS and 18F]-fluorocholine PET / CT in the assessment of metabolism of the choline. To establish the diagnosis value of both methods, separately and in combination.
* To determine which examinations are useful and complementary for the diagnosis and the management of gliomes.

FET combined with MRS may be a powerful, widely applicable new method to improve the diagnosis of cerebral gliomas. The extent to which FCH and MRS provide similar information is not known precisely and this study will establish their respective diagnostic value in differentiating tumoral from non-tumoral tissue.

ELIGIBILITY:
Inclusion Criteria:

* Suspicion of intracerebral glioma on MR
* Men of women
* Age >18, no upper limit as long as a biopsy or intervention is foreseen

Exclusion Criteria:

* Need of rapid intervention in <2 weeks
* Previous neurosurgical intervention (biopsy, shunt, etc.) or any other cerebral treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with glioma suspicion referred for biopsy to our university hospital
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2009-07; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Ability of image-guided biopsy using FET, FCH PET/CT and MRS information to target the most representative sites of tumor grade as compared to histopathological examination | On the biopsy day

CONTACTS AND LOCATIONS:
Overall Officials: John O Prior, PhD MD, Principal Investigator — Centre Hospitalier Universitaire Vaudois and University of Lausanne
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Lausanne, CH, Switzerland

IPD SHARING:
Plan to Share IPD: No